CLINICAL TRIAL: NCT00877162
Title: Night Waking Reduction in Canadian Infants: A Randomized Controlled Clinical Trial of a Parent-based Cognitive and Behavioural Intervention in Community Health Units.
Brief Title: The Rocky Sleep Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H09-00757; CIHR MCT-94836
Record Dates: First submitted 2009-04-03; First posted 2009-04-07 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Sleep Problems
Keywords: Cognitive and behavioural intervention; trial; group; Behavioral sleep problems
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Providing parents with a group teaching intervention (2 hours long). The teaching session is followed by 2 weeks of phone calls twice a week to offer parents support for their use of the strategies described in the teaching session and to clarify any questions about the teaching session content. The arm will have baseline data collected one week prior to the teaching session. Follow-up data will be collected at 6 and 24 weeks post intervention. A pamphlet on infant safety will be distributed to the intervention arm following the 6 week data collection point. A pamphlet on managing behavioural sleep problems will distributed to the control group following the 6 week data collection point.
  Interventions: Behavioral: Controlled crying and routines

INTERVENTIONS:
Behavioral: Controlled crying and routines — Behavioural (teaching and support)

SUMMARY:
Night waking with crying can be a distressing and difficult experience for infants and their parents. The investigators want to reduce infant night waking and crying and improve parents' views of their infants' sleep. This study will help the investigators determine whether parents who receive group teaching about infant sleep and follow-up phone calls provided by Public Health Nurses will reduce numbers of infants' night wakes and parents' perceptions of infant sleep difficulties compared with parents who receive a group teaching about infant safety and follow-up phone calls provided by Public Health Nurses. Results from this study will help the investigators improve their practice when assisting parents and infants with sleep problems.

DETAILED DESCRIPTION:
Background: Infant behavioural sleep problems affect up to 50% of infants, can persist, and can contribute to adverse developmental outcomes. Persistent short night sleep periods from 5-to 29 months of age have been associated with more hyperactivity and inattention, and lower abilities at cognitive tasks for older children. Sleep problems in infants are also associated with parental stress, fatigue and family tension, and maternal depression. Health care professionals often fail to recognize and treat infant sleep problems and over 40 books and many websites provide conflicting advice. Interventions directed at changing parents' cognitions and behaviours have reduced infant night waking and reduced parents' distress; however, inexpensive, short term group interventions to improve infant sleep problems and reduce effects of conflicting advice are needed. Parents' knowledge about infant sleep affects their behaviours at bedtime and responses to night waking. Combined cognitive-behavioural approaches can modify those factors and improve outcomes.

Research Design: The study is a randomized controlled trial aimed at 6 to 8-month-old infants who are waking at night and crying, with stratification by community health centres and blinded analysis of actigraphic/sleep diary data Primary Question: In a population of parents who have infants with behavioural sleep problems are parents randomized to a cognitive-behavioural sleep intervention compared to parents randomized to a group cognitive-behavioural safety intervention more or less likely to: a) identify their child as having a severe sleep problem, or b) to have their child wake fewer than an average of 2 times per night over 5 nights by actigraphy? Inclusion criteria: Biological or adoptive parents who: 1) read and speak English, 2) have access to a telephone, and 3) are in two parent or single parent families. Infants who are: 1) healthy, 2) between 5.5 and 8 months of age, and 3) screened and identified as having a sleep problem.

Exclusion criteria: Infants with: 1) organic causes of sleep disruption, 2) developmental disability, and 3) chronic neurological or respiratory conditions. Parents with 1) diagnosed depression, 2) diagnosed sleep problems, and 3) permanent night shift work.

Sample size: The team will randomize 240 families with infants to the control or experimental group.

The Intervention: We will recruit families through programs at community 5 health centres, the Vancouver Coastal Health Website, and the Newborn Hotline. Prior to randomization, experimental and control groups will be screened for infant sleep problems and provide baseline data by questionnaire (sleep cognitions, depression, sleep quality, and fatigue), infant sleep diaries and actigraphy. The intervention has high ecological validity, because public health nurses will offer a group format with 1 teaching session and four phone calls in a community setting. The experimental group and control group will receive a short 2 hour teaching session to change cognitions and behaviour to manage infant sleep problems and infant safety respectively. For the experimental group, cognitions include thoughts about normal infant sleep and developmental appropriateness of infant self-soothing. Both groups will receive two weeks of telephone support twice weekly.

Primary Outcome: A significant infant sleep disturbance as measured with a composite measure, which will consist of either parent reporting a severe sleep problem OR mean actigraphic wakes of greater than 2 per night averaged over 5 nights at 6 weeks post-teaching session. The control group will receive a sleep pamphlet after 6 weeks and experimental group will receive a safety pamphlet.

Analysis: All analysis will follow the intent-to-treat principle. We will apply Fisher's exact test to compare outcome prevalence of our primary composite of severe problems or wakes averaging more than 2 per night over 5 nights between groups. We will assess variation between health units using logistic regression, incorporating terms for health unit and health unit by treatment interaction.

Significance: The trial will be complete in 30 months and has the potential to build capacity in community health nurses to offer systematic programs to manage infant sleep problems.

ELIGIBILITY:
Inclusion Criteria:

* Parents and their healthy 5.5 to 8 month-old infants.
* Infants are waking 2 or more times per night or more than 20 minutes for at least 4 nights per week for a minimum of 3 weeks.
* Parents are biological or have adopted their infants, can speak and read English, have access to a telephone and are in two or one parent families.

Exclusion Criteria:

* Infants are excluded who have biological causes of sleep problems, developmental disability, and/or chronic neurological or respiratory conditions.
* Parents are excluded who have diagnosed depression and are receiving treatment, have diagnosed sleep problems (e.g. sleep apnea), and are working permanent night shifts.

Ages: 6 Months to 8 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 235 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Severity of infant sleep problem on a severity scale (parents' perception) | 6 & 24 weeks

SECONDARY OUTCOMES:
Less than an average of twice a night over 5 nights by actigraphy | 6 & 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Hall, RN, PhD, Principal Investigator — University of British Columbia; Radhika Bhagat, RN, MN, Study Director — Vancouver Coastal Health; Rollin Brant, Ph.D, Study Director — Centre for Community Child Health Research; Jean Paul Collett, Ph.D, Study Director — Child and Family Research Institute; Amiram Gafni, Ph.D, Study Director — McMaster University; Dorothy Hamilton, RN, BSN, Study Director — Vancouver Coastal Health; Eileen Hutton, Ph.D, Study Director — McMaster University; Kathy Hydamaka, RN, BSN, Study Director — Vancouver Coastal Health; Osman Ipsiroglu, MD, Study Director — Sunny Hill Health Centre for Children; Valerie Munroe, RN, MSN, Study Director — Vancouver Coastal Health Research Institute; Roy Saunders, MD, Study Director — Seymour Medical Clinic; Kathy Triolet, RN, BSN, Study Director — Vancouver Coastal Health; Lillian Tse, RN, MSN, Study Director — Vancouver Coastal Health; Joanne Wooldridge, RN, MSN, Study Director — Vancouver Coastal Health
Locations (5):
- Canada (5):
  - Richmond Community Health Services, Richmond, British Columbia
  - North Shore Coastal Community Health, Vancouver, British Columbia
  - Pacific Spirit Community Health Centre, Vancouver, British Columbia
  - South Community Health Office, Vancouver, British Columbia
  - Three Bridges Community Health Centre, Vancouver, British Columbia

REFERENCES:
- [Derived] Hall WA, Hutton E, Brant RF, Collet JP, Gregg K, Saunders R, Ipsiroglu O, Gafni A, Triolet K, Tse L, Bhagat R, Wooldridge J. A randomized controlled trial of an intervention for infants' behavioral sleep problems. BMC Pediatr. 2015 Nov 13;15:181. doi: 10.1186/s12887-015-0492-7. PMID 26567090